CLINICAL TRIAL: NCT01586143
Title: Clinical Study Comparing the Efficacy of Transbuccal Paracetamol 125 mg Versus Paracetamol Injection 1g in Slow Infusion IV in Patients With Acute Pain
Acronym: PARAJUG
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CHU-0118
Record Dates: First submitted 2012-04-10; First posted 2012-04-26 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Acute Pain
Keywords: Paracetamol by permucosal route,; Paracetamol by intraveinous route,; Pain.; Patient with minor trauma of lower limb and/or superior limb (sprains, muscle contusions, …).
MeSH Terms: conditions — Acute Pain; Pain; Sprains and Strains | interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider

ARMS (2):
- transbuccal paracetamol 125 mg (Experimental): This is a clinical study that aims to investigate and compare the efficacy of transbuccal paracetamol 125 mg with that of paracetamol 1g administered intravenously in patients with acute pain of moderate intensity accepted to emergency room following a minor trauma of the lower limbs and/or superiors. To this end, several pain scoring will be performed using a visual analogue scale (VAS) at various times after drug administration.
  Interventions: Drug: paracetamol
- placebo (Placebo Comparator): This is a clinical study that aims to investigate and compare the efficacy of transbuccal paracetamol 125 mg with that of paracetamol 1g administered intravenously in patients with acute pain of moderate intensity accepted to emergency room following a minor trauma of the lower limbs and/or superiors. To this end, several pain scoring will be performed using a visual analogue scale (VAS) at various times after drug administration.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: paracetamol — This is a clinical study that aims to investigate and compare the efficacy of transbuccal paracetamol 125 mg with that of paracetamol 1g administered intravenously in patients with acute pain of moderate intensity accepted to emergency room following a minor trauma of the lower limbs and/or superiors. To this end, several pain scoring will be performed using a visual analogue scale (VAS) at various times after drug administration.
  Arms: transbuccal paracetamol 125 mg
Drug: Placebo
  Arms: placebo

SUMMARY:
This is a clinical study that aims to investigate and compare the efficacy of transbuccal paracetamol 125 mg with that of paracetamol 1g administered intravenously in patients with acute pain of moderate intensity accepted to emergency room following a minor trauma of the lower limbs and/or superiors. To this end, several pain scoring will be performed using a visual analogue scale (VAS) at various times after drug administration.

DETAILED DESCRIPTION:
This is a clinical study that aims to investigate and compare the efficacy of transbuccal paracetamol 125 mg with that of paracetamol 1g administered intravenously in patients with acute pain of moderate intensity accepted to emergency room following a minor trauma of the lower limbs and/or superiors. To this end, several pain scoring will be performed using a visual analogue scale (VAS) at various times after drug administration.

ELIGIBILITY:
Inclusion Criteria:

* Patient admitted to emergency departments with trauma of upper or lower limbs (sprains, muscle contusions,…) associated with intensity moderate of acute pain (VAS between 4 and 6) which require infusion IV of paracetamol 1g.
* Patient takes any chronic treatment which considered incompatible with study.
* Patient between 18 and 60.
* Male or female.
* Sufficient cooperation and understanding to comply to the requirements of study.
* Acceptance to give a written consent.
* Affiliation at system of French social security.
* Inscription or acceptation of inscription at national register of voluntaries participant at research

Exclusion Criteria:

* Against paracetamol-indication: hypersensitivity known at paracétamol, antecedent hepatitis B or C, severe renal insufficiency and liver failure.
* Patient with medical or surgical antecedents.
* Patient with progressive disease at balance of inclusion.
* Alcoholism suspicion or toxicomany at intake.
* Patient who presents any inflammation or ulcerative pathology about buccal mucosa.
* Patient who refuses to ingest alcohol for personal reasons.
* Woman in childbearing age not using effective contraceptive method, pregnant or lactating woman.
* Patient who participated in another clinical trial, located in exclusion period or received benefits > 4500 euros during 12 months before the beginning of trial.
* Patient with cooperation and understanding insufficiency to comply to the requirements of protocol
* Patient with social protection
* No affiliation at system of French social security

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2012-05; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Pain score measured by visual analogue scale | at T0 + 120 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Gisele PICKERING, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Derived] Pickering G, Moustafa F, Macian N, Schmidt J, Pereira B, Dubray C. A New Transmucous-Buccal Formulation of Acetaminophen for Acute Traumatic Pain: A Non-inferiority, Randomized, Double-Blind, Clinical Trial. Pain Physician. 2015 May-Jun;18(3):249-57. PMID 26000668